CLINICAL TRIAL: NCT00347880
Title: Atrial and Brain Natriuretic Peptides in Bronchiolitis
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB# 359-2004; GCRC 602
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; ANP; BNP; Atrial Natriuretic Peptide; Brain Natriuretic Peptide; Vasopressin; ADH; Pediatric; Respiratory Distress; Fluid Balance
MeSH Terms: conditions — Bronchiolitis; Diabetes Insipidus; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to collect information about what happens to certain chemicals produced in the body called hormones during respiratory infections such as bronchiolitis. Bronchiolitis is an infection of small airways in the lungs caused by a virus. This infection, which causes swelling and injury in the lungs, is commonly seen in infants and children less than 2 years of age.

DETAILED DESCRIPTION:
Intravascular volume and serum osmolality are tightly regulated by a balance of various neurohumoral mediators. In critical illness, these regulatory mediators may be modified by disease or treatment, either benefiting or harming the patient. Such regulatory mediators of intravascular volume and fluid balance include atrial natriuretic peptide (ANP), brain natriuretic peptide (BNP) and vasopressin (also called antidiuretic hormone-ADH). Although well studied in adult cardiac patients, these neurohormones have not been investigated in pediatric respiratory diseases such as bronchiolitis, a common cause of admission to the Pediatric Intensive Care Unit (PICU). Understanding the effects of pediatric respiratory diseases and treatment interventions on the concentrations of these neurohormonal regulators such as ANP and BNP is a crucial first step in formulating more effective fluid therapy. For example, some patients with bronchiolitis have elevated ADH levels. Increased ADH concentration predisposes to fluid retention and increases the risk of pulmonary edema. Since ANP and BNP antagonize the action of ADH, simultaneous measurement of all three hormones may help elucidate the mechanisms of fluid balance in bronchiolitis.

The study hypothesis is that the plasma concentrations of ANP and BNP in infants and children with bronchiolitis are inversely associated with ADH concentration and lung hyperinflation. Furthermore, plasma concentrations of ANP and BNP in bronchiolitis are associated directly with increased oxygen requirement and positive fluid balance. The significance of this study is to better understand the relationship between various neurohormones that regulate intravascular fluid volume in patients with respiratory failure and bronchiolitis. The understanding of this complex relationship has the potential to improve fluid/diuretic therapy and patient outcome with severe respiratory distress in the future.

We plan to enroll 100 patients in this study. The population will be infants and children between 37 weeks and 2 years of age (corrected for gestational age). 50 patients with bronchiolitis will be enrolled to collect ANP, BNP, and ADH plasma levels along with serum osmolality and urine osmolality for up to 5 consecutive days in Shands Children's Hospital.

Comparison: 50 control patients will be enrolled to record normal baseline plasma ANP, BNP, and ADH at the time of admission in Shands Hospital surgical center at the University of Florida.

ELIGIBILITY:
Inclusion Criteria:

* child between 37 weeks and 2 years old
* chest X-ray evidence of peri-bronchial cuffing or air trapping
* Two of the Following:
* history or evidence of nasal secretion
* inter-and/or sub-costal retractions
* evidence of wheezing

Exclusion Criteria:

* acute or chronic renal disease
* chronic diuretic therapy
* congenital cardiac disease
* bronchopulmonary dysplasia
* thyroid disease
* pituitary abnormalities
* history of reactive airway disease
* asthma
* cystic fibrosis
* recent history of receiving steroids

Ages: 37 Weeks to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between the ages of 37 weeks and 2 years old with evidence of bronchiolitis.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2004-09; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K. Alex Daneshmand, D.O., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States